CLINICAL TRIAL: NCT02068989
Title: Stress Hyperglycemia as an Indicator for Future Diabetes Mellitus: A Prospective Cohort Study
Brief Title: Study of Stress Hyperglycemia as an Indicator of Diabetes Mellitus
Status: Terminated | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 1301011408
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Stress Hyperglycemia; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stress Hyperglycemic Group: Repeat HbA1C in 1 year
- Euglycemic Group: Repeat HbA1C in 1 year

SUMMARY:
We hypothesize that stress hyperglycemia is an indicator that a patient will develop type 2 diabetes mellitus in the future. Subjects who are not diabetic are enrolled and blood glucose readings reviewed during their intensive care unit stay. All subjects are consented and have a HbA1C level drawn to determine if they have diabetes mellitus or not. They are then followed up in 1 year and the HbA1C repeated to determine if they have developed diabetes mellitus over the course.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intensive care unit at the Yale New Haven Hospital St. Raphael Campus and Norwalk Hospital

Exclusion Criteria:

* Patients with prior history of diabetes mellitus
* Elevated admission HbA1c (≥6.5%)
* Age >80 years
* Metastatic disease with expected life expectancy of less than 12 months
* Pregnancy or a woman who plans to become pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit admissions who are not known to be diabetic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Subjects with an HbA1c greater than or equal to 6.5% | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Atlas, MD, Principal Investigator — Yale New Haven Hospital; Jonathon Fine, MD, Principal Investigator — Norwalk Hospital
Locations (2):
- United States (2):
  - Yale New Haven Hospital St. Raphael Campus, New Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut